CLINICAL TRIAL: NCT04667923
Title: Noninvasive Ventilation in Moderate-to-severe COVID-19-associated Acute Respiratory Distress-syndrome to Prevent Tracheal Intubation: the COVID-NIV Study
Brief Title: Noninvasive Ventilation in Moderate-to-severe COVID-19-associated Acute Respiratory Distress-syndrome
Acronym: COVID-NIV
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 002-NIV-COVID
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2020-12

CONDITIONS: Covid19; ARDS
MeSH Terms: conditions — COVID-19 | interventions — Capnography; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Respiratory monitoring — Measurement of the tidal volume, peak inspiratory flow, inspiratory time, respiratory rate and the pressure gap during triggering on NIV and plateau pressure on mechanical ventilation
Diagnostic Test: Respiratory muscles ultrasound — Measurement of the diaphragm thickening fraction, assessment of the contraction of scalene and sternocleidomastoid muscles
Diagnostic Test: Electro impedance tomography — Measurement of the lung impedance changes in 4 quadrants, measurement of regional ventilation delay in 4 quadrants
Diagnostic Test: Capnography — Measurement of end-tidal carbon dioxide tension
Diagnostic Test: Arterial blood gas — Measurement of the oxygen partial pressure and the carbon dioxide partial pressure
Diagnostic Test: Quasistatic pressure-volume curve — Quasistatic pressure-volume curve

SUMMARY:
Non-invasive ventilation can allow to avoid intubation and improve outcomes in moderate-to-severe COVID-19-associated acute respiratory distress-syndrome (ARDS). Data on NIV parameters adjustment based on expanded respiratory and gas exchange monitoring in COVID-19 associated ARDS is limited. Appropriate adjustment of the inspiratory positive airway pressure (IPAP) set as a point of the balance between minimal work of breathing (minimum point of W.Patrick scale for assessment of the accessory respiratory muscles and minimum diaphragm thickening fraction) and minimum tidal volume, and respiratory rate can decrease NIV failure in moderate-to-severe COVID-ARDS. The objective of the study is to evaluate the ability of non-invasive ventilation guided with expanded respiratory monitoring to decrease the intubation rate in in moderate-to-severe COVID-ARDS.

DETAILED DESCRIPTION:
In December 2019, an outbreak of a novel coronavirus emerged in Wuhan, China and rapidly spread worldwide. The World Health Organization (WHO) declared the outbreak a pandemic on March 11th, 2020. The clinical disease (COVID-19) results in critical illness in about 5% of patients with predominant acute respiratory failure.

The objective of the study is to evaluate the ability of non-invasive ventilation guided with expanded respiratory monitoring to decrease the intubation rate in in moderate-to-severe COVID-ARDS. Investigators will set IPAP as a point of the balance between minimal work of breathing (minimum point of W.Patrick scale for assessment of the accessory respiratory muscles, and minimum diaphragm thickening fraction) and minimum tidal volume, and respiratory rate. Investigators will set expiratory pressure at 8-10 cm of water and the inspiratory oxygen fraction (FiO2) to reach oxygen saturation by pulse oximetry (SpO2) 95%. All gas exchange measurements will be set at IPAP level. For gas exchange assessment investigators will measure partial oxygen tension in the arterial blood (PaO2), partial carbon dioxide tension in arterial blood (PaCO2), end-tidal carbon dioxide tension (PetCO2), then will calculate PAO2/FiO2, alveolar dead space (Vd alv) and ventilatory ratio (VR). Investigators will measure expiratory tidal volume (VT), respiratory rate (RR), peak inspiratory flow (PIF) and inspiratory time at 3 levels: at the set IPAP, at IPAP+4 cm of water and at IPAP-4 cm of water. Measurements will be repeated on day 1, 3, 5, 7, 14 and 21 of NIV. NIV failure is determined as one of the following at set IPAP 26 cm of water and FiO2 100%: fatigue, Patrick scale 5 points, SpO2<92%, apnoea, hemodynamic instability or Glasgow coma score <14 points.

In patients with NIV failure after intubation and every 7 day after intubation investigators will measure plateau pressure and calculate the driving pressure at PEEP 8-10-12-14 cm of water and VT 6 ml/kg predicted body weight (PBW), and VT+100 ml and VT+200 ml at PEEP 8 cm of water, plot static pressure volume-curve at positive end-expiratory pressure (PEEP) 5 and 14 cm of water, and perform electro impedance tomography.

This study is an observational trial in the ICU of the University hospital.

ELIGIBILITY:
Inclusion Criteria:

* at least one of the following criteria: fatigue, Patrick scale 5 points, SpO2<92% on standard oxygen therapy (<15 l/min) or continuous positive airway pressure (CPAP)-therapy with oxygen flow<15 l/min

Exclusion Criteria:

* pregnancy
* age less than 18 or more than 80 years
* life-threatening heart rhythm abnormalities and/or systolic blood pressure < 80 mmHg despite norepinephrine at a dose > 2 µg/kg/min
* primary lung diseases (e.g. interstitial lung diseases, lung emphysema) or tumour metastases in lungs
* chronic decompensated diseases with extrapulmonary organ dysfunction (tumour progression, liver cirrhosis, congestive heart failure)
* Glasgow cona score < 14
* inability to swallow
* upper airways obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with COVID-19-associated moderate-to-severe acute respiratory distress-syndrome
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Intubation rate | On day 28
  Frequency of NIV failure
Mortality | On day 28
  Mortality on day 28

SECONDARY OUTCOMES:
Change in arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio | Days 1, 3, 5, 7, 10, 14, 21 during noninvasive ventilation
  Calculation of the arterial partial oxygen tension to inspiratory oxygen fraction (PaO2/FiO2) ratio using arterial oxygen tension measurement
Change in ventilatory ratio | Days 1, 3, 5, 7, 10, 14, 21 during noninvasive ventilation
  Measurement of arterial carbon dioxide tension, minute ventilation and calculation of ventilatory ratio
Change in alveolar dead space | Days 1, 3, 5, 7, 10, 14, 21 during noninvasive ventilation
  Calculation of the alveolar dead space using end-tidal carbon dioxide measurement and arterial carbon dioxide tension measurement
Change in tidal volume | Days 1, 3, 5, 7, 10, 14, 21 during noninvasive ventilation
  Measurement of exhaled tidal volume
Change in accessory respiratory muscles workload | Days 1, 3, 5, 7, 10, 14, 21 during noninvasive ventilation
  Calculation of the Patrick's scale (minimum 0 points, maximum 5 points, more points means worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey I Yaroshetskiy, MD, PhD, ScD, Principal Investigator — Sechenov University
Locations (1):
- Sechenov University clinic #4, Moscow, Russia

REFERENCES:
- [Background] Avdeev SN, Yaroshetskiy AI, Tsareva NA, Merzhoeva ZM, Trushenko NV, Nekludova GV, Chikina SY. Noninvasive ventilation for acute hypoxemic respiratory failure in patients with COVID-19. Am J Emerg Med. 2021 Jan;39:154-157. doi: 10.1016/j.ajem.2020.09.075. Epub 2020 Oct 1. PMID 33067061
- [Background] Agarwal R, Handa A, Aggarwal AN, Gupta D, Behera D. Outcomes of noninvasive ventilation in acute hypoxemic respiratory failure in a respiratory intensive care unit in north India. Respir Care. 2009 Dec;54(12):1679-87. PMID 19961634
- [Background] Yaroshetskiy AI, Avdeev SN, Konanykhin VD. Acute Respiratory Distress Syndrome in COVID-19: Do All These Patients Definitely Require Intubation and Mechanical Ventilation? Am J Respir Crit Care Med. 2020 Nov 15;202(10):1480-1481. doi: 10.1164/rccm.202007-2713LE. No abstract available. PMID 32809841
- [Background] Patrick W, Webster K, Ludwig L, Roberts D, Wiebe P, Younes M. Noninvasive positive-pressure ventilation in acute respiratory distress without prior chronic respiratory failure. Am J Respir Crit Care Med. 1996 Mar;153(3):1005-11. doi: 10.1164/ajrccm.153.3.8630538.
- [Derived] Yaroshetskiy AI, Merzhoeva ZM, Tsareva NA, Trushenko NV, Nuralieva GS, Konanykhin VD, Krasnoshchekova AP, Avdeev SN. Breathing pattern, accessory respiratory muscles work, and gas exchange evaluation for prediction of NIV failure in moderate-to-severe COVID-19-associated ARDS after deterioration of respiratory failure outside ICU: the COVID-NIV observational study. BMC Anesthesiol. 2022 Oct 1;22(1):307. doi: 10.1186/s12871-022-01847-7. PMID 36183064